CLINICAL TRIAL: NCT01647932
Title: Safety and Efficacy of the Combination of Loop Diuretics With Thiazide-type Diuretics in Patients With Decompensated Heart Failure: a Double-blind, Randomized, Placebo-controlled Trial (CLOROTIC Trial).
Brief Title: Safety and Efficacy of the Combination of Loop With Thiazide-type Diuretics in Patients With Decompensated Heart Failure
Acronym: CLOROTIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Society of Internal Medicine (Other)
Responsible Party: Principal Investigator, Joan Carles Trullas Vila, Principal Investigator, Spanish Society of Internal Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEMI-IC-CLOR
Record Dates: First submitted 2012-06-28; First posted 2012-07-24 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Diuretics; Diuretic resistance
MeSH Terms: conditions — Heart Failure | interventions — Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loop plus thiazide-type diuretic (Active Comparator): Loop diuretic plus hydrochlorothiazide
  Interventions: Drug: hydrochlorothiazide
- Loop diuretic plus placebo (Placebo Comparator): Loop diuretic plus placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hydrochlorothiazide — hydrochlorothiazide according to clearance of creatinine; >50ml/min 25mg daily, 20-50ml/min 50mg daily amd <20ml/min 100mg daily.
  Arms: Loop plus thiazide-type diuretic
Drug: Placebo — Placebo according to clearance of creatinine; >50ml/min 1/2 pill daily, 20-50ml/min 1 pill daily amd <20ml/min 2 pills daily.
  Arms: Loop diuretic plus placebo

SUMMARY:
The purpose of this study is to determine whether a combined diuretic therapy (loop diuretics with thiazide-type diuretics) is more effective (in terms of improving fluid overload symptoms) among patients with decompensated heart failure in comparison with loop diuretic alone.

DETAILED DESCRIPTION:
Volume overload is an important clinical target in heart failure management, typically addressed using loop diuretics. An important and challenging subset of heart failure patients exhibit fluid overload despite significant doses of loop diuretics. One approach to overcome loop diuretic resistance is the addition of a thiazide-type diuretic to produce diuretic synergy via "sequential nephron blockade," first described more than 40 years ago. Although potentially able to induce diuresis in patients otherwise resistant to high doses of loop diuretics, this strategy has not been subjected to large-scale clinical trials to establish safety and clinical efficacy. Combination diuretic therapy using any of several thiazide-type diuretics can more than double daily urine sodium excretion to induce weight loss and edema resolution. To our knowledge there are no clinical trials designed to prove the efficacy and safety of combined diuretic therapy (a commonly used therapy) among patients with decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic heart failure
* Admission for acute decompensated heart failure
* There is no prespecified inclusion criterion with respect to heart failure etiology and/or ejection fraction
* Receipt of an oral loop diuretic for at least 1 month before hospitalization, at a dose between 80 mg and 240 mg daily in the case of furosemide and an equivalent dose in the case of a different loop diuretic (20 mg of torasemide or 1 mg of bumetanide was considered to be equivalent to 40 mg of furosemide)

Exclusion Criteria:

* Other etiologies of fluid overload different from heart failure
* Hyponatremia: any symptomatic sodium value or a sodium level below 125mmol/l
* Unstable patients: acute coronary syndrome, cardiogenic shock or ICU admission.
* Patients requiring inotropic agents or renal replacement therapies
* Life expectancy < 6 months
* Prior treatment with thiazide-type diuretics
* Aldosterone antagonists are permitted if the patient had been taking them on a long-term basis (at least 30 days before randomisation)
* Pregnancy or breastfeeding period
* Active alcoholism and/or other substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2014-10; Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | Bodyweight will be measured every 24 hours (during hospitalisation) from the date of inclusion / randomisation until the date of discharge.
  Bodyweight will be measured every 24 hours (during hospitalisation) from the date of inclusion / randomisation until the date of discharge.
  Changes in body weight measurements: the mean of weight lost every 24 hours and the total weight lost from baseline to the 5th day of hospitalisation.
  Participants will be followed for the duration of hospital stay, an expected average of 9 days.
Patient-reported dyspnea | Patient-reported dyspnea is assessed every 24 hours (during hospitalisation) from the date of inclusion / randomisation until the date of discharge.
  Patient-reported dyspnea is assessed every 24 hours (during hospitalisation) from the date of inclusion / randomisation until the date of discharge.
  Patient-reported dyspnea is assessed with the use of a visual-analogue scale (VAS) and the Linker 7 point scale.
  Changes in patient-reported dyspnea: changes in the dyspnea scales from baseline to the 5th day of hospitalisation.

SECONDARY OUTCOMES:
Diuresis | 24-hour diuresis will be quantified every 24 hours (during hospitalisation) from the 1st day until the 4th day of hospitalisation.
Worsening renal function | Renal function will be determined every 24 hours (during hospitalisation) from the date of inclusion / randomisation until the date of discharge.
  Renal function will be determined every 24 hours (during hospitalisation) from the date of inclusion / randomisation until the date of discharge.
  Renal function is assessed with the serum creatinine level. Worsening renal function is defined as an increase in the serum creatinine level of more than 0.3 mg/dl at any time during hospitalisation Participants will be followed for the duration of hospital stay, an expected average of 9 days.
Changes in electrolyte levels (sodium and potassium) | Electrolyte levels (sodium and potassium) will be determined every 24 hours (during hospitalisation) from the date of inclusion / randomisation until the date of discharge.
  Electrolyte levels (sodium and potassium) will be determined every 24 hours (during hospitalisation) from the date of inclusion / randomisation until the date of discharge.
  Electrolyte levels are assessed with the serum sodium and potassium levels. Participants will be followed for the duration of hospital stay, an expected average of 9 days.
Metrics of diuretic response | weight loss and net fluid loss per mg of furosemide
  weight loss and net fluid loss per mg of furosemide
Mortality (all-cause and heart failure) | Mortality (all-cause and heart failure) at 30 and 90days post-discharge
  Mortality (all-cause and heart failure) at 30 and 90days post-discharge
Rehospitalization (all-cause and heart failure) | Rehospitalization (all-cause and heart failure) at 30 and 90days post-discharge
  Rehospitalization (all-cause and heart failure) at 30 and 90days post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Joan Carles Trullas, MD, PhD, Principal Investigator — Heart Failure Study Group, Spanish Society of Internal Medicine
Locations (1):
- Internal Medicine Service, Hospital d'Olot (Girona), Olot, Girona, Spain

REFERENCES:
- [Background] Jentzer JC, DeWald TA, Hernandez AF. Combination of loop diuretics with thiazide-type diuretics in heart failure. J Am Coll Cardiol. 2010 Nov 2;56(19):1527-34. doi: 10.1016/j.jacc.2010.06.034. PMID 21029871
- [Background] ter Maaten JM, Valente MA, Damman K, Hillege HL, Navis G, Voors AA. Diuretic response in acute heart failure-pathophysiology, evaluation, and therapy. Nat Rev Cardiol. 2015 Mar;12(3):184-92. doi: 10.1038/nrcardio.2014.215. Epub 2015 Jan 6. PMID 25560378
- [Background] Trullas JC, Morales-Rull JL, Casado J, Freitas Ramirez A, Manzano L, Formiga F; CLOROTIC investigators. Rationale and Design of the "Safety and Efficacy of the Combination of Loop with Thiazide-type Diuretics in Patients with Decompensated Heart Failure (CLOROTIC) Trial:" A Double-Blind, Randomized, Placebo-Controlled Study to Determine the Effect of Combined Diuretic Therapy (Loop Diuretics With Thiazide-Type Diuretics) Among Patients With Decompensated Heart Failure. J Card Fail. 2016 Jul;22(7):529-36. doi: 10.1016/j.cardfail.2015.11.003. Epub 2015 Nov 11. PMID 26576715
- [Background] Trullas JC, Morales-Rull JL, Formiga F. [Diuretic therapy in acute heart failure]. Med Clin (Barc). 2014 Mar;142 Suppl 1:36-41. doi: 10.1016/S0025-7753(14)70081-8. Spanish. PMID 24930082
- [Background] Trullas JC, Casado J, Morales-Rull JL, Formiga F, Conde-Martel A, Quiros R, Epelde F, Gonzalez-Franco A, Manzano L, Montero-Perez-Barquero M. Prevalence and outcome of diuretic resistance in heart failure. Intern Emerg Med. 2019 Jun;14(4):529-537. doi: 10.1007/s11739-018-02019-7. Epub 2019 Jan 4. PMID 30610440
- [Derived] Conde-Martel A, Hernandez-Meneses M, Morales-Rull JL, Casado J, Carrera-Izquierdo M, Leon M, Sanchez-Marteles M, Davila-Ramos MF, Hernandez-Carballo C, Llacer P, Moreno-Garcia MC, Salamanca-Bautista P, Formiga F, Manzano L, Trullas JC. Hypokalemia During Decongestion With Loop Diuretics and Hydrochlorothiazide, a Post Hoc Analysis of the CLOROTIC Trial. Circ Heart Fail. 2025 Sep;18(9):e012914. doi: 10.1161/CIRCHEARTFAILURE.125.012914. Epub 2025 Jul 1. PMID 40590131
- [Derived] Conde-Martel A, Trullas JC, Morales-Rull JL, Casado J, Carrera-Izquierdo M, Sanchez-Marteles M, Llacer P, Salamanca-Bautista P, Manzano L, Formiga F. Sex differences in clinical characteristics and outcomes in the CLOROTIC (combining loop with thiazide diuretics for decompensated heart failure) trial. Rev Clin Esp (Barc). 2024 Feb;224(2):67-76. doi: 10.1016/j.rceng.2023.11.003. Epub 2024 Jan 11. PMID 38215973
- [Derived] Trullas JC, Morales-Rull JL, Casado J, Carrera-Izquierdo M, Sanchez-Marteles M, Conde-Martel A, Davila-Ramos MF, Llacer P, Salamanca-Bautista P, Chivite D, Jordana-Comajuncosa R, Villalonga M, Paez-Rubio MI, Manzano L, Formiga F. Combining loop and thiazide diuretics for acute heart failure across the estimated glomerular filtration rate spectrum: A post-hoc analysis of the CLOROTIC trial. Eur J Heart Fail. 2023 Oct;25(10):1784-1793. doi: 10.1002/ejhf.2988. Epub 2023 Aug 16. PMID 37540036
- [Derived] Trullas JC, Morales-Rull JL, Casado J, Carrera-Izquierdo M, Sanchez-Marteles M, Conde-Martel A, Davila-Ramos MF, Llacer P, Salamanca-Bautista P, Perez-Silvestre J, Plasin MA, Cerqueiro JM, Gil P, Formiga F, Manzano L; CLOROTIC trial investigators. Combining loop with thiazide diuretics for decompensated heart failure: the CLOROTIC trial. Eur Heart J. 2023 Feb 1;44(5):411-421. doi: 10.1093/eurheartj/ehac689. PMID 36423214